CLINICAL TRIAL: NCT01499849
Title: Phase 3, Multicenter, Randomized, Double Blind, Active-Controlled Study of the Safety & Efficacy of Rolapitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Subjects Receiving Highly Emetogenic Chemotherapy (HEC)
Brief Title: Ph3 Safety/Efficacy Study of Rolapitant for the Prevention of CINV in Subjects Receiving Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TS-P04832
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2012-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Rolapitant; Nausea; Vomiting; CINV; Chemotherapy
MeSH Terms: conditions — Vomiting; Nausea | interventions — rolapitant; Granisetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rolapitant (Experimental): Day 1: Rolapitant (200 mg PO) + Granisetron (10 mcg/kg IV) + dexamethasone (20 mg PO) Days 2-4: Dexamethasone (8 mg PO) will be administered orally BID.
  Interventions: Drug: Rolapitant; Drug: Granisetron; Drug: dexamethasone
- Placebo + Granisetron + Dexamethasone (Placebo Comparator): Day 1: Placebo + Granisetron (10 mcg/kg IV)+ dexamethasone (20 mg PO) Days 2-4: Dexamethasone (8 mg PO) will be administered orally BID.
  Interventions: Drug: Granisetron; Drug: dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Rolapitant — (4 X 50 mg capsules) 200 mg PO
  Other Names: Varubi
  Arms: Rolapitant
Drug: Granisetron — 10 mcg/kg IV
  Other Names: Kytril; Granisol
Drug: dexamethasone — 20 mg PO and 8 mg PO
  Other Names: Decadron
Drug: Placebo — (4 X 0 mg capsules) 0 mg PO
  Other Names: Placebo to match Rolapitant
  Arms: Placebo + Granisetron + Dexamethasone

SUMMARY:
This is a Phase 3, multicenter, randomized, parallel-group, double-blind, active-controlled study of rolapitant in subjects receiving HEC. Rolapitant or placebo will be administered prior to initiation of chemotherapy on Day 1 with granisetron and dexamethasone. Subjects will record all events of emesis and use of rescue medication for established nausea and/or vomiting, and will indicate the severity of nausea they experienced in each of the previous 24 hours in the Nausea and Vomiting (NV) Subject Diary prior to HEC administration through Day 6 of Cycle 1. Health-related quality of life will be measured by the FLIE Questionnaire on Day 6 of Cycle 1. Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examinations, electrocardiograms (ECGs), and safety laboratory values.

All subjects are expected to complete Cycle 1 and will have the option of participating in up to five additional cycles.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, parallel-group, double-blind, active-controlled study of rolapitant in subjects receiving HEC (≥60 mg/m2 of cisplatin-based chemotherapy). Study drug will be administered 1 - 2 hours prior to initiation of chemotherapy on Day 1. Granisetron and dexamethasone will be administered approximately 30 minutes before initiation of chemotherapy on Day 1,except in patients receiving taxanes as part of cisplatin-based chemotherapy. Subjects will record all events of emesis and use of rescue medication for established nausea and/or vomiting and will indicate the severity of nausea they experienced in each of the previous 24 hours in the NV Subject Diary prior to HEC administration through Day 6 in Cycle 1. Dexamethasone 8 mg twice daily (part of study regimen) on Days 2 through 4 is NOT considered rescue therapy. Health-related quality of life will be measured by the FLIE Questionnaire on Day 6 of Cycle 1. Safety and tolerability will be assessed by clinical review of AEs, physical examinations including complete neurological assessment, vital signs,electrocardiograms (ECGs), and safety laboratory values including BUN andcreatinine. All subjects are expected to complete Cycle 1 and will have the option of participating in up to five additional cycles. The study will investigate the efficacy of rolapitant for the treatment of CINV during an initial chemotherapy cycle (Cycle 1).

Safety analyses will include data from Cycle 1 and from subsequent cycles. At the Screening Visit, blood samples may be collected and stored in this study and maybe analyzed for future biomarker research related to safety and efficacy. Analysis of these samples may include DNA, RNA, or protein markers. The biomarker blood samples will be stored for up to 2 years post study completion. In addition, PK samples will be collected from subjects enrolled in selected sites.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, of either gender, and of any race
* has never been treated with cisplatin and is to receive the first course of cisplatin-based chemotherapy (≥60 mg/m2)
* Karnofsky performance score of ≥60
* Predicted life expectancy of ≥4 months
* Adequate bone marrow, kidney, and liver function

Exclusion Criteria:

* Contraindication to cisplatin, granisetron, or dexamethasone
* Is pregnant or breast feeding
* Has previously received cisplatin or subject is planning to receive multiple days of cisplatin in a single cycle
* Has taken the following agents within the last 48 hours 5-HT3 antagonists,Phenothiazines,Benzamides,Domperidone,Cannabinoids,NK1 antagonist, Benzodiazepines
* Scheduled to receive any other chemotherapeutic agent with an emetogenicity level of 4 or above (Hesketh Scale) from Day 2 through Day 6, except on Day 1.
* Scheduled to receive any radiation therapy to the abdomen or pelvis from Day -5 through Day 6
* Has received systemic corticosteroids or sedative antihistamines within 72 hours of Day 1 of the study except as premedication for chemotherapy (e.g., taxanes, pemetrexed)
* symptomatic primary or metastatic CNS disease.
* Has ongoing vomiting, retching, clinically significant nausea caused by any etiology, or has a history of anticipatory nausea and vomiting.
* Has vomited and/or has had dry heaves/retching within 24 hours prior to the start of cisplatin-based chemotherapy on Day 1 in Cycle 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — Tesaro, Inc.
Locations (1):
- TESARO Inc, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Rapoport BL, Chasen MR, Gridelli C, Urban L, Modiano MR, Schnadig ID, Poma A, Arora S, Kansra V, Schwartzberg LS, Navari RM. Safety and efficacy of rolapitant for prevention of chemotherapy-induced nausea and vomiting after administration of cisplatin-based highly emetogenic chemotherapy in patients with cancer: two randomised, active-controlled, double-blind, phase 3 trials. Lancet Oncol. 2015 Sep;16(9):1079-1089. doi: 10.1016/S1470-2045(15)00035-2. Epub 2015 Aug 10. PMID 26272769

RESULTS

PARTICIPANT FLOW:
Groups:
- Rolapitant + Granisetron + Dexamethasone: * Oral dose of rolapitant 180 mg (equivalent to 200 mg rolapitant hydrochloride monohydrate) 1-2 h before administration of chemotherapy
  * Granisetron (10 μg/kg intravenously) about 30 min before chemotherapy
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy, and dexamethasone 8 mg orally twice daily on days 2-4
- Placebo + Granisetron + Dexamethasone: * Matching placebo 1-2 h before administration of chemotherapy
  * Granisetron (10 μg/kg intravenously) about 30 min before chemotherapy
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy, and dexamethasone 8 mg orally twice daily on days 2-4
Period: Overall Study
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Started | 266 (Number of randomized patients) | 266
Completed | 42 (Number of patients who completed 6 cycles) | 40
Not Completed | 224 | 226
Not completed — Adverse Event | 28 | 32
Not completed — Chemo completed or Change in Therapy | 70 | 67
Not completed — Withdrawal by Subject | 43 | 43
Not completed — Death | 5 | 7
Not completed — Disease Progression | 11 | 10
Not completed — Protocol Violation | 11 | 11
Not completed — Physician Decision | 20 | 19
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 6 | 3
Not completed — Other Reasons | 27 | 30

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants only included the Modified Intent to Treat (MITT) population:
  * 266 subjects were randomized to Rolapitant and 266 were randomized to control;
  * 264 of those randomized to Rolapitant received study drug in Cycle 1; 262 of those who were randomized to control received study drug in Cycle 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone | Total
Number analyzed (Participants) | 264 | 262 | 526
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.08) | 57.7 (11.15) | 57.3 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 112 | 222
  Male | 154 | 150 | 304
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 34 | 67
  Not Hispanic or Latino | 231 | 228 | 459
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 61 | 56 | 117
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 178 | 179 | 357
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: No Emetic Episodes and No Rescue Medication
Description: The primary objective of this study is to determine whether administration of rolapitant with granisetron and dexamethasone improves CINV in the delayed phase (>24 to 120 hours) of CINV compared with administration of placebo with granisetron and dexamethasone in subjects receiving HEC. The primary outcome will be based on complete response (defined as no emetic episodes and no rescue medication) in the delayed phase (>24 to 120 hours).
Time Frame: >24 to 120 hours post chemotherapy
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 264 | 262
percentage of participants | 72.7 [66.9 to 78.0] | 58.4 [52.2 to 64.4]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. For the CR delayed the threshold for statistical significance was 0.05; no further adjustment for multiplicity were required for the primary endpoint; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.3 to 2.7]

2. Secondary Outcome: Acute Phase Response
Description: To determine the effect of rolapitant on complete response rates in the acute (0 to 24 hours)phase of CINV
Time Frame: 0 to 24 hours
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 264 | 262
percentage of participants | 83.7 [78.7 to 88.0] | 73.7 [67.9 to 78.9]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. CR-acute was tested only if the result for the primary endpoint, CR delayed, was statistically significant; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.2 to 2.8]

3. Secondary Outcome: Overall Response Rate
Description: To determine the effect of rolapitant on complete response rates in the overall (0 to 120 hours) phase of CINV.
Time Frame: 0 to 120 hours
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 264 | 262
percentage of participants | 70.1 [64.2 to 75.5] | 56.5 [50.2 to 62.6]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. CR overall was tested only if both CR delayed and CR acute were statistically significant; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.3 to 2.6]

ADVERSE EVENTS:
Time Frame: Up to 6 cycles of treatment (median number cycles=2; median duration of each cycle = 21-22 days)
Description: Safety analysis was based on actual treatment received in Cycle 1. 266 subjects were randomized to Rolapitant, among which 263 received Rolapitant in Cycle 1, hence Safety=263 for Rolapitant. 266 subjects were randomized to control, among which 263 received control in Cycle 1 (There was an error in treatment received), hence Safety=263 for control.
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 37/263 | 54/263
Other Adverse Events (participants affected / at risk) | 187/263 | 198/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rolapitant + Granisetron + Dexamethasone (N=263) | Placebo + Granisetron + Dexamethasone (N=263)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Impaired Gastric Empyting (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 3
Disease Progression (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Multi-Organ Failure (General disorders) | 0 | 2
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1
Bronchitis Bacterial (Infections and infestations) | 1 | 0
Encephalitis Herpes (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infective Exacerabation of Bronchiectasis (Infections and infestations) | 0 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Septic Shock (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Stromal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 1 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 2
Loss of Consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rolapitant + Granisetron + Dexamethasone (N=263) | Placebo + Granisetron + Dexamethasone (N=263)
Anaemia (Blood and lymphatic system disorders) | 28 | 32
Leukopenia (Blood and lymphatic system disorders) | 18 | 14
Neutropenia (Blood and lymphatic system disorders) | 33 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 12
Constipation (Gastrointestinal disorders) | 26 | 29
Diarrhoea (Gastrointestinal disorders) | 20 | 18
Dyspepsia (Gastrointestinal disorders) | 18 | 8
Nausea (Gastrointestinal disorders) | 24 | 35
Stomatitis (Gastrointestinal disorders) | 16 | 14
vomiting (Gastrointestinal disorders) | 9 | 22
Asthenia (General disorders) | 35 | 40
Fatigue (General disorders) | 36 | 30
Mucosal Inflammation (General disorders) | 17 | 19
Decreased Appetite (Metabolism and nutrition disorders) | 30 | 36
Dehydration (Metabolism and nutrition disorders) | 13 | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No